CLINICAL TRIAL: NCT07376434
Title: The Relationship Between Sexual Health Literacy and Artificial Intelligence Literacy in Young Adults: A Cross-Sectional Digital Age Study
Brief Title: Sexual Health and Artificial Intelligence Literacy in Young Adults: Digital Age Perspective
Status: Recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Eslem Altıntaş, MSc, Acibadem University
Other Study IDs: 2026-01/3
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Sexuality; Artificial Intelligence
Keywords: Young Adults; Sexuality; Artificial Intelligence
MeSH Terms: conditions — Sexuality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young Adults Participants: Participants aged 18-24 years, able to read and write Turkish, with internet access, voluntarily participating in this observational cross-sectional study.

SUMMARY:
Young people represent a substantial proportion of the global population, and the experiences gained during adolescence and early adulthood play a critical role in shaping lifelong health behaviors. Health literacy, defined as the ability to access, understand, and use health information, is particularly important during this developmental period.

Sexual health is a key component of overall well-being and quality of life. Risky sexual behaviors among young adults may lead to serious outcomes such as unintended pregnancies, sexually transmitted infections, and sexual violence. Therefore, sexual health literacy is essential for promoting safe behaviors and protecting reproductive health.

In recent years, digital environments have become major sources of health information for young people. With the rapid rise of generative artificial intelligence tools, individuals increasingly rely on AI-based systems for accessing and interpreting health-related content. This highlights the growing importance of artificial intelligence literacy, which refers to the ability to understand, critically evaluate, and effectively use AI technologies.

However, the relationship between artificial intelligence literacy and sexual health literacy has not yet been directly examined. This study aims to investigate the association between these two literacy domains among young adults, contributing to a better understanding of sexual health information-seeking behaviors in the digital age.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-24 years
* Able to read and write Turkish
* Access to the internet
* Voluntarily agreeing to participate

Exclusion Criteria:

* Refusal to provide informed consent
* Visual impairment preventing survey completion
* Cognitive or language impairments preventing survey completion

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of young adults aged 18-24 years living in Turkey. Participants are recruited online via social media and digital communication channels. Only those who can read and write Turkish, have internet access, and voluntarily agree to participate are included.
Sampling Method: Non-Probability Sample
Enrollment: 269 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Introduction Information Forum | At enrollment
  This form was developed by the researchers based on the relevant literature and consists of 29 items designed to assess participants' sociodemographic characteristics and digital usage patterns.
Sexual Health Literacy | At enrollment (18-24 years old participants)
  Sexual health literacy assessed using the 17-item Sexual Health Literacy Scale. The scale includes two subscales: Knowledge (12 items, score range 12-60) and Attitude (5 reverse-coded items, score range 5-25). Higher scores indicate higher sexual health literacy. Cronbach's alpha = 0.88.
Artificial Intelligence Literacy | At enrollment (18-24 years old participants)
  AI literacy assessed using the 12-item Artificial Intelligence Literacy scale, covering four dimensions: Awareness, Usage, Evaluation, Ethics. Each item scored 1-5; higher scores indicate greater AI literacy. Cronbach's alpha = 0.939.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Coşkun, Ph.D., Principal Investigator — Acibadem University; Güzin Ünlü Suvari, M.Sc., Principal Investigator — Acibadem University
Locations (1):
- Online study, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Üstgörül, S. (2022). Development of a sexual health literacy scale: Validity and reliability study. Ankara Journal of Health Sciences, 11(2), 164-176.
- [Background] Broder J, Okan O, Bauer U, Bruland D, Schlupp S, Bollweg TM, Saboga-Nunes L, Bond E, Sorensen K, Bitzer EM, Jordan S, Domanska O, Firnges C, Carvalho GS, Bittlingmayer UH, Levin-Zamir D, Pelikan J, Sahrai D, Lenz A, Wahl P, Thomas M, Kessl F, Pinheiro P. Health literacy in childhood and youth: a systematic review of definitions and models. BMC Public Health. 2017 Apr 26;17(1):361. doi: 10.1186/s12889-017-4267-y. PMID 28441934